CLINICAL TRIAL: NCT02883400
Title: Spironolactone to Prevent or Delay Calcineurin Inhibitor (CNI) Toxicity in Liver Transplant Recipients
Brief Title: Spironolactone After Liver Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-14-03A
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2021-06

CONDITIONS: Transplant, Liver
MeSH Terms: interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOC-Standard of care (No Intervention): standard of care, nontreatment
- spironolactone (Experimental): spironolactone
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — spironolactone 25 mg up to 50 mg
  Arms: spironolactone

SUMMARY:
To study spironolactone to prevent calcineurin inhibitor (CNI) kidney injury.

DETAILED DESCRIPTION:
The aim of this study is to determine if spironolactone decreases nephrotoxicity from calcineurin inhibitors in liver transplant recipients and to determine the best study of renal function in liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* liver transplant

Exclusion Criteria:

* dual organ transplant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark W. Russo, MD, MPH, Principal Investigator — Charolinas Healthcare System
Locations (1):
- CHS, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Russo MW, Krista Bossi, Gale Groseclose, Levi DM, Lon Eskind, Bennett Noell, Anderson WE, Zamor PJ, Vincent Casingal. Estimates of Glomerular filtration rate in liver transplant recipients are not accurate: A role for 24 hour urine creatinine clearance. Archives of Transplantation 2018:2:1-5.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SOC-Standard of Care | Spironolactone
Started | 22 | 8
Completed | 22 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOC-Standard of Care | Spironolactone | Total
Number analyzed (Participants) | 22 | 8 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 8 | 27
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Full Range); unit: years] | 55 [23 to 70] | 55 [39 to 64] | 55 [23 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 19 | 5 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 19 | 8 | 27
  Black or African American | 1 | 0 | 1
  Hispanic or Latino | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 22 | 8 | 30
Glomerular Filtration Rate [Mean (Inter-Quartile Range); unit: mL/min//1.73m^2] | 90 [50 to 110] | 90 [54 to 110] | 90 [50 to 110]

OUTCOME MEASURES:

1. Primary Outcome: Glomerular Filtration Rate (GFR)
Description: The primary analyses were based on the difference between each estimated GFR measure and iothalamate scan.
Time Frame: 18 months
Population: liver transplant recipients
Measure: Mean (Inter-Quartile Range); unit: ml/min/1.73m^2
Groups:
- SOC-Standard of Care: Standard of care
- Spironolactone: spironolactone group
Arm/Group | SOC-Standard of Care | Spironolactone
Number analyzed (Participants) | 22 | 8
ml/min/1.73m^2 | 69 [50 to 110] | 64 [54 to 110]
Statistical Analysis 1: Comparison: SOC-Standard of Care vs Spironolactone; Test type: Superiority; p = 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 5

ADVERSE EVENTS:
Time Frame: 18 months
Description: adverse events were collected according to clinical trials. gov defintions or by clinical descrption
Arm/Group | SOC-Standard of Care | Spironolactone
All-Cause Mortality (participants affected / at risk) | 0/22 | 1/8
Serious Adverse Events (participants affected / at risk) | 2/22 | 2/8
Other Adverse Events (participants affected / at risk) | 1/22 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC-Standard of Care (N=22) | Spironolactone (N=8)
Fever (General disorders) | 2 (2) | 2 (2) — 2 patients in SOC arm and 2 patients in treatment arm were hospitalized for Fever.
cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 1 (1) — Subject expired from cardiopulmonary arrest and liver failure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC-Standard of Care (N=22) | Spironolactone (N=8)
elevated serum potassium (Blood and lymphatic system disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT02883400/Prot_SAP_000.pdf